CLINICAL TRIAL: NCT01859104
Title: Feasibility and Efficacy of Engagement Modules for Renal and Liver Transplant Candidates
Brief Title: Feasibility of Use of BariCare App in Pre-transplant Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: App to be used in study needs revision.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Manpreet S. Mundi, Assistant Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-001535
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Pre-Renal Transplant Candidate; Pre-liver Transplant Candidate
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smartphone Arm (Other): This is a feasibility trial and thus all participants in the study will be provided a smartphone app to assist them in making lifestyle modifications
  Interventions: Behavioral: Use of smartphone app

INTERVENTIONS:
Behavioral: Use of smartphone app

SUMMARY:
This current study aims to evaluate the efficacy of engagement modules in assisting patients who are candidates for renal and liver transplantation make significant lifestyle modifications. With the help of the Center for Innovation (CFI), a smartphone app (Android and iOS compatible) has been created to assist in both educating and engaging patients to develop and maintain healthy lifestyle modifications. Our goal is to create a cost-effective, smartphone-based platform that serves to not only efficiently educate but to also verify competence and keep our patients engaged.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are candidates for liver or renal transplant.
2. Individuals who own a smartphone.
3. Individuals who are obese.

Exclusion Criteria:

1. Patients with prior history of bariatric surgery.
2. Patients with active psychiatric disorder.
3. Patients with active tobacco use.
4. Patients with active substance use (alcohol, illicit drugs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Smart Phone App Feasibility | 3 months
  The primary objective will be to assess ease and feasibility of use by subjects. They will provide information through questionnaires developed to assess these factors.

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet Mundi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided